CLINICAL TRIAL: NCT05470192
Title: The Effects of Qigong Exercise Training on Shoulder and Respiratory Function After Thoracotomy
Brief Title: The Effects of Qigong Exercise Training After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Neriman Temel Aksu, Research Assistant (Expert Physiotherapist), Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AU
Record Dates: First submitted 2022-06-30; First posted 2022-07-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Pain, Shoulder; Postoperative Pain; Joint Adhesion; Muscle Weakness; Respiratory Function Loss; Quality of Life
Keywords: Thoracotomy; Qigong exercise training; Shoulder function; Respiratory function; Quality of life; Pain
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Muscle Weakness; Respiratory Aspiration; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Exercise Training and Conventional Physiotherapy and Rehabilitation Group (Experimental): In addition to the conventional physiotherapy and rehabilitation program, qigong exercise training will be given to the qigong exercise training group by a certified physiotherapist who has received qigong training.
  Interventions: Other: Qigong exercise training
- Conventional Physiotherapy and Rehabilitation Group (No Intervention): A training will be given including information about the postoperative recovery process, the purpose of respiratory physiotherapy and rehabilitation, the importance of physiotherapy and rehabilitation in the postoperative period, attention to speed up recovery and prevention of complications, breathing exercises, coughing training, posture exercises, early mobilization and its importance, and answering patient questions. . The program includes progressive ambulation and progressive shoulder and rib cage exercises. These exercises will be performed under the supervision of a physiotherapist from the first postoperative day. The exercises will be advanced every day by increasing the number of repetitions.

INTERVENTIONS:
Other: Qigong exercise training — Before and after the qigong exercises, 10-minute exercises will be done to stretch the large muscle groups for warm-up-cooling purposes.
  The entire Baduanjin exercise consists of 8 postures:
  preparation position
  1. Raising arms with palms up,
  2. Shooting arrows left and right like an archer in a semi-crouching position
  3. Keeping one arm up
  4. Looking back with trunk rotations in a semi-crouching position
  5. Nodding the head and lowering the body to relieve stress,
  6. Fisting and staring
  7. Touching feet with hands touching back and legs
  8. Raising and lowering heels
  Other Names: Therapeutic Baduanjin Qigong Exercises
  Arms: Qigong Exercise Training and Conventional Physiotherapy and Rehabilitation Group

SUMMARY:
Postoperative pulmonary complications after thoracotomy cause morbidity and mortality. Although the causes of postoperative pulmonary complication are multifactorial, respiratory muscle dysfunction is a contributing factor to the development of postoperative pulmonary complication. This phenomenon has been explained by changes in respiratory muscle mechanics and operative function. Exercise interventions following lung resection have been shown to be associated with benefits on functional capacity, quality of life, shoulder pain, and shoulder function. Following thoracotomy, postoperative pulmonary complications are a significant cause of morbidity and cause significant increase in health care costs, intensive care and hospital stay, and patient discomfort. Conventional physiotherapy and rehabilitation program applied after thoracotomy reduces hospital stay and incidence of atelectasis.

Thoracotomy may also result in long-term limitation of shoulder function and range of motion, reduced muscle strength, chronic pain, and reduced health-related quality of life. Physiotherapy program; It provides some benefits such as reduction of pain, improvement of shoulder function and physical components of quality of life. Based on these findings; It is recommended that physiotherapists provide a postoperative exercise program aimed at reducing shoulder dysfunction and pain, including progressive shoulder and rib cage exercises and a home program after discharge.

In recent years, the popularity of Tai Chi, Qigong and yoga, also known as body-mind exercises in the treatment of chronic diseases, has increased.

DETAILED DESCRIPTION:
A standard posterolateral thoracotomy incision is usually performed in lung surgery due to its various advantages. Standard posterolateral thoracotomy is also used in lung problems such as lung parenchyma problems, hydatid cyst, mesothelioma, bullous disease of the lung along with cancer. In a standard posterolateral thoracotomy, the latissimus dorsi and serratus anterior muscles are cut. Latissimus dorsi muscle; Although it is very effective in deep inspiration, strong cough, shoulder girdle activity, it is also the accessory muscle of expiration. When the past 90 years are examined, standard posterolateral thoracotomy; It has been found that there are some disadvantages such as postoperative pulmonary complications due to cutting large muscle groups, increased potential blood loss, restricted shoulder and upper extremity joint range of motion, prolonged dysfunction, scoliosis formation, severe and chronic postoperative pain and cosmetic problems. These; Cutting large muscle groups, damaging the shoulder girdle muscles, restricting shoulder and upper extremity joint movements, causing postoperative pulmonary failure, pain and morbidity. The standard posterolateral thoracotomy is the most commonly used incision in non-cardiac open thoracic surgical procedures. The fact that it can be applied in all thoracic pathologies makes it the most used incision. Allowing the operating surgeon and assistant to use their hands together in the thoracic cavity and providing a good view for the thoracic cavity; posterolateral thoracotomy is the advantages of the incision.

Postoperative pulmonary complications after thoracotomy cause morbidity and mortality. Although the causes of postoperative pulmonary complication are multifactorial, respiratory muscle dysfunction is a contributing factor to the development of postoperative pulmonary complication. This phenomenon has been explained by changes in respiratory muscle mechanics and operative function. Exercise interventions following lung resection have been shown to be associated with benefits on functional capacity, quality of life, shoulder pain, and shoulder function. Physiotherapy interventions have been used regularly since the 1960s for the prevention and treatment of both pulmonary and musculoskeletal complications following major surgery. Following thoracotomy, postoperative pulmonary complications are a significant cause of morbidity and cause significant increase in health care costs, intensive care and hospital stay, and patient discomfort. Conventional physiotherapy and rehabilitation program applied after thoracotomy reduces hospital stay and incidence of atelectasis. Early postoperative pulmonary rehabilitation after lung surgery can improve lung function by increasing cardiopulmonary and peripheral muscle endurance of patients.

Thoracotomy can also cause long-term limitation of shoulder function and range of motion, reduced muscle strength, chronic pain, and reduced health-related quality of life. Physiotherapy program; It provides some benefits such as reduction of pain, improvement of shoulder function and physical components of quality of life. Based on these findings; It is recommended that physiotherapists provide a postoperative exercise program aimed at reducing shoulder dysfunction and pain, including progressive shoulder and rib cage exercises and a home program after discharge.

In a study, it was found that a postoperative exercise program accompanied by a physiotherapist provides significant benefits in pain and shoulder functions for patients after open thoracotomy. During the hospital stay, physiotherapists focus on the prevention and management of postoperative pulmonary complications and the improvement of patients' thoracic and shoulder mobility. Among the treatment methods for postoperative pulmonary complications; breathing exercises consisting of active breathing technique, deep breathing exercises, incentive spirometry, continuous maximum inspiration, intermittent positive pressure breathing and positive expiratory pressure devices, cough maneuvers and forced expiratory technique. In addition, early-stage functional activities such as getting out of bed, taking steps in place, walking, climbing stairs and cycling have been included as treatment options for postoperative pulmonary complications and to improve physical function. Maintaining shoulder and trunk mobility can be achieved with shoulder and trunk range of motion exercises.

In recent years, the popularity of Tai Chi, Qigong and yoga, also known as body-mind exercises in the treatment of chronic diseases, has increased.

They are recommended as a category of exercise that includes a range of movements and body positions, focused on breathing, defined by a calm state of mind and deep relaxation. These exercises are; It includes many common components such as mind-focused, slow, relaxed, fluent, respiratory-oriented, and providing deep physical and mental relaxation.

Tai Chi and Qigong exercises are rooted in ancient China, as are traditional Chinese medicine practices. Originally a spiritual practice, Yoga originated in India. These practices have been shown to have many health benefits. Many randomized controlled trials such as fibromyalgia, breast cancer, cardiovascular conditions, and diabetes have focused on the positive effects of moving meditation on specific medical conditions of various populations.

In addition to conventional physiotherapy and rehabilitation after thoracotomy, Qigong exercise training applied for 8 weeks; In this study, which was planned to evaluate the effects on shoulder function, shoulder joint range of motion, shoulder muscle strength, post-thoracotomy incision pain and shoulder pain, dyspnea respiratory function, respiratory muscle strength, functional capacity and quality of life, he was hospitalized in Akdeniz University Hospital Thoracic Surgery clinic and underwent standard posterolateral thoracotomy. Patients who meet the criteria between 20-70 years of age will be taken. The control group will consist of patients who received conventional physiotherapy and rehabilitation in the post-thoracotomy period. The study group, on the other hand, will consist of patients who underwent qigong exercises in addition to the conventional physiotherapy and rehabilitation program in the post-thoracotomy period.

Pain, shoulder mobility, shoulder muscle strength, shoulder function, dyspnea, respiratory function, respiratory muscle strength, respiratory muscle endurance, functional capacity, quality of life will be evaluated for outcome measures.

Evaluations will be repeated in the preoperative period, postoperative 7th day, postoperative 4th week, and postoperative 8th week.

Conventional physiotherapy and rehabilitation will be applied to all patients participating in the study.

The program includes progressive ambulation and progressive shoulder and rib cage exercises. These exercises will be performed under the supervision of a physiotherapist from the first postoperative day.

The exercises will be advanced every day by increasing the number of repetitions. In addition to the study group, 8 weeks of Qigong exercise training will be applied.

As a result of the literature study, no study was found that evaluated the effectiveness of qigong exercise training applied after thoracotomy on shoulder and respiratory functions. Therefore, in our study; qigong exercise training to be applied in addition to conventional physiotherapy after thoracotomy; It is thought that it will reduce shoulder and upper extremity joint range of motion, limitation in shoulder functions, decrease in shoulder muscle strength, postoperative pulmonary complications, and increase quality of life and functions.

The hypotheses of the study are as follows. H0: Shoulder and respiratory functions of the patients who underwent qigong exercise training after thoracotomy were not better than the control group.

H1: Shoulder and respiratory functions of the patients who underwent qigong exercise training after thoracotomy were better than the control group.

This study will be performed on patients who will undergo posterolateral thoracotomy surgery in the Department of Thoracic Surgery of Akdeniz University Medical Faculty Hospital. The control group will consist of patients who underwent conventional physiotherapy and rehabilitation in the post-thoracotomy period. The study group will consist of patients who underwent qigong exercises in addition to the conventional physiotherapy and rehabilitation program in the post-thoracotomy period.

ELIGIBILITY:
Inclusion Criteria:

* Posterolateral thoracotomy surgery
* Hemodynamically stable
* Who agreed to participate in the study

Exclusion Criteria:

* Decortication, undergoing thoracic wall surgery
* Patients with known cerebrovascular disease and related neurologic involvement
* Using any device for ambulation
* Those who have undergone shoulder surgery within 6 months
* Those with cognitive dysfunction (Mini Mental Test score <24)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change of Pain Score | Change from Baseline Pain Score at 8 weeks.
  The person is asked to rate their pain between 0 and 10 (0=Absence of Pain, 10=The Most Unbearable Pain). Numerical Pain Rating Scale is frequently used because of its ease of use. The scale can be completed in 1 minute. Three pain regions will be evaluated in this study. These regions; the incision line (along the incision or within the two intercostal spaces above or below), over the rib cage (outside the incision site), and the shoulder joint complex (upper extremity and trapezius muscle near the middle humerus, including the clavicular and scapular areas). They will be asked to score and indicate numerically between 0 and 10 points. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Active Shoulder Range of Motion | Change from Baseline Active Shoulder Range of Motion at 8 weeks.
  Active shoulder range of motion of the patients will be evaluated with a digital goniometer (Baseline Digital Absolute & Axis Goniometer) using a standard protocol. Total shoulder motion that allows motion of all joints in the shoulder complex will be measured, glenohumeral motion will not be isolated. Flexion, abduction, external and internal rotation of the shoulder will be evaluated. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Shoulder Muscle Strength | Change from Baseline Shoulder Muscle Strength at 8 weeks.
  Shoulder muscle strength will be measured using a dynamometer (MicroFET 2 Manual Muscle Tester). Force measurements will be taken for shoulder flexion, abduction, internal and external rotation. Before starting the test, patients will be informed about how to perform the test. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Pulmonary Function | Change from Baseline Pulmonary Function at 8 weeks.
  The Pulmonary Function Test will be performed with the COSMED Pony FX (COSMED; Italy) spirometer in accordance with the criteria of the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Forced vital capacity (FVC), Forced expiratory volume in 1 second (FEV1), Tiffeneau ratio (FEV1/FVC), Forced expiratory flow 25-75% (FEF25-75%) and peak expiratory flow rate (PEF) values and predictive values percentage will be recorded. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Respiratory Muscle Strength | Change from Baseline Respiratory Muscle Strength at 8 weeks.
  Respiratory muscle strength measurement will be performed with a portable, electronic intraoral pressure measuring device COSMED Pony FX (COSMED; Italy) according to ATS/ERS criteria. The MIP will be measured at residual volume and during deep inspiration. MEP will be determined at total lung capacity and during deep expiration. Measurements will be made in a sitting position using a nose clip. Patients will be verbally encouraged for the best strength. Measurement will be made until it provides the valid value in patients. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Respiratory Muscle Endurance | Change from Baseline Respiratory Muscle Endurance at 8 weeks.
  Respiratory Muscle Endurance will be performed by COSMED Pony FX (COSMED; Italy) spirometry by applying the maximal voluntary ventilation (MVV) procedure in accordance with the criteria of the American Thoracic Society (ATS) and the European Respiratory Society (ERS). The patient will be asked to breathe deeper and faster than the resting tidal volume for 12 seconds. When the test is finished after 12 seconds, the device will show the predictive value of MVV % that we used in our study. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Functional Capacities | Change from Baseline Functional Capacities at 8 weeks.
  The functional capacities of the patients will be measured with the 6-minute walking test. Before testing, patients will rest for 10 minutes. Before starting the test, patients should be told if they feel too short of breath during the test; It will be explained that they can slow down, stop and rest, and this time will be included in the test. Patients will be asked to walk as fast as possible at their own walking pace for 6 minutes on a 30-meter straight corridor. Fatigue and dyspnea perception will be assessed with the Modified Borg Scale. The Modified Borg Scale was developed to measure the effort spent during exercise and is a scale that is frequently used to evaluate the severity of exertional dyspnea and the severity of dyspnea at rest. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Basal Dyspnea Index Score | Change from Baseline of Basal Dyspnea Index Score at 8 weeks.
  Basal Dyspnea Index will be applied to evaluate the dyspnea status of the patients. Basal Dyspnea Index (Baseline Dyspnea Index, BDI): BDI is a scale developed to evaluate dyspnea due to activity. Its Turkish validity and reliability have been established by different researchers. The scale consists of three sub-dimensions: functional status (level of performing activities of daily living), effort capacity (difficult efforts to perform activities), and work capacity. Each sub-dimension is scored between 0 (very severe impairment) and 4 (no impairment). The total score ranges from 0 to 12, and as the score decreases, the severity of dyspnea increases. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Quality of Life Score | Change from Baseline Quality of Life Score at 8 weeks.
  The quality of life of our patients will be evaluated using the Short Form-12. Health-related quality of life refers to the function and well-being of the physical, mental and social dimensions of life. SF-12 are among the most used multi-element health-related quality-of-life instruments. Preoperative period, postoperative 4th week and postoperative 8th week will be repeated.
Change of Shoulder, Pain and Disability Index Score | Change from Baseline Shoulder, Pain and Disability Index Score at 8 weeks.
  Shoulder function will be measured using the Shoulder, Pain and Disability Index , a self-rated questionnaire designed to measure shoulder pain and disability. Shoulder Pain and Disability Index is a reliable questionnaire evaluating shoulder pain and disability. Turkish reliability and validity were performed by Bumin et al. in 2008. There are 2 subscales and 13 items in total in the index. 5 of them evaluate pain and 8 evaluate disability. The items of both subscales are measured with a visual analog scale from 0 to 10. The scores given by the individual are added together and calculated as a percentage. Higher scores indicate more severe pain and higher disability. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated

SECONDARY OUTCOMES:
Height in Meters | Initial assessment before surgery
  The height of all subjects in meters (m) will be noted before the surgery.
Weight in Kilograms | Initial assessment before surgery
  The weight of all subjects in kilograms (kg) will be noted before the surgery.
Body Mass Index (BMI) in kg/m^2 | Initial assessment before surgery
  Body Mass Index (BMI) will be calculated with the formula weight (kg)/height (m)^2.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman T Aksu, Principal Investigator — Akdeniz Üniversitesi
Locations (1):
- Neriman Temel Aksu, Antalya, Turkey (Türkiye)